CLINICAL TRIAL: NCT02294097
Title: The Outcomes of Protocol-Specified Modification of Immunosuppression Directed to Histological Diagnosis by Surveillance Protocol Biopsy
Brief Title: Protocol-Specified Modification of Immunosuppression Directed to Protocol Biopsy in Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wiwat Chancharoenthana, Chulalongkorn University, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WWC-005
Record Dates: First submitted 2014-11-15; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Surveillance Protocol Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-biopsy (No Intervention): Population in this arm will be adjusted immunosuppressive drug only from the result of tough level.
- Protocol biopsy (Experimental): Population in this arm will be adjusted immunosuppressive drug upon both pathological findings and the result of tough level.
  Interventions: Procedure: Surveillance protocol kidney allograft biopsy

INTERVENTIONS:
Procedure: Surveillance protocol kidney allograft biopsy — Surveillance protocol biopsy under ultrasound-guided will perform at post-operative day 7, month 3, month 6, month 12, and month 24
  Arms: Protocol biopsy

SUMMARY:
The risk-benefit of surveillance-protocol biopsy (SPBx) in kidney transplantation remains unclear. The study aims to compare outcomes of recipients with SPBx approach to recipients with standard approach which allograft biopsy was performed only when indicated.

DETAILED DESCRIPTION:
The present randomized-controlled trial in kidney transplant patients aims to compare the outcomes and complications between who underwent immunosuppessive drug modification under surveillance-protocol biopsy and who underwent immunosuppressive drug modification following tough level only.

ELIGIBILITY:
Inclusion Criteria:

* All kidney transplant recipients underwent transplantation at Chulalongkorn University

Exclusion Criteria:

* Pregnancy
* Recipients who cannot withhold aspirin, clopidogrel, warfarin, etc.
* Non-cooperated recipients

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Renal function | 24 months
  24 h-CrCl

SECONDARY OUTCOMES:
Renal pathology | 24 months
  interstitial fibrosis, rejection, calcineurin inhibitor toxicity
Complications | immediate, 1 month
  hematoma, arteriovenous fistula

CONTACTS AND LOCATIONS:
Overall Officials: Wiwat Chancharoenthana, MD.,MSc., Principal Investigator — Chulalongkorn University
Locations (1):
- Division of Nephrology, Department of Medicine, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand